CLINICAL TRIAL: NCT06134934
Title: TeleCare North Diabetes: A Feasibility Study
Brief Title: TeleCare North Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Steno Diabetes Center Nordjylland (Other); Aalborg University (Other)
Responsible Party: Principal Investigator, Peter Vestergaard, MD, professor, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N-20230026
Record Dates: First submitted 2023-11-01; First posted 2023-11-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Blood glucose; Diabetes mellitus; Type 2; Telemedicine; Telehealth; Telemonitoring; Feasibility
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telemonitoring design 1 (Experimental): * Self-Monitoring of Blood Glucose (SMBG)
  * Sleep
  * Mental health
  * Blood pressure
  * Activity
  Interventions: Other: Telemonitoring 1
- Telemonitoring design 2 (Experimental): * Self-Monitoring of Blood Glucose (SMBG)
  * Sleep
  * Mental health
  Interventions: Other: Telemonitoring 2

INTERVENTIONS:
Other: Telemonitoring 1 — This telemonitoring intervention design include self-monitoring of blood glucose (SMBG) together with monitoring of sleep, mental health, blood pressure and activity.
  Arms: Telemonitoring design 1
Other: Telemonitoring 2 — This telemonitoring intervention design include self-monitoring of blood glucose (SMBG) together with monitoring of sleep and mental health.
  Arms: Telemonitoring design 2

SUMMARY:
This feasibility study will evaluate the feasibility of two telemonitoring designs for non-insulin treated T2D patients with an eye to identify the most suitable telemonitoring intervention for a future large-scale randomized trial.

DETAILED DESCRIPTION:
Background: Maintaining optimal glycaemic control in type 2 diabetes (T2D) is difficult. Telemedicine has potential to support poorly controlled people with T2D in the achievement of glycaemic control if the telemedicine solution includes a telemonitoring component. However, only few telemonitoring solutions for non-insulin treated T2D exist. Therefore, the aim of this feasibility study is to evaluate the feasibility of two telemonitoring intervention designs for non-insulin treated T2D patients with an eye to identify the most suitable telemonitoring intervention for a future large-scale randomized trial.

Method: The trial will be conducted as a three-month randomized feasibility study in four municipalities in North Denmark with 15 participants from each municipality. Two different telemonitoring intervention designs will be tested. One intervention will include self-monitoring of blood glucose (SMBG) together with monitoring of sleep and mental health. The second intervention will include an identical setup but with the addition of blood pressure and activity monitoring. Two municipalities will be allocated to one intervention design, whereas the other two municipalities will be allocated to the second intervention design. Qualitative interviews with participants and clinicians will be conducted to gain insight into their experiences with and acceptance of the intervention designs and trial procedures (e.g., blood sampling and questionnaires). In addition, differences in direct intervention costs between the two alternative interventions will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women and men ≥ 18 years
* Poorly controlled T2D, i.e. HbA1c > 58 mmol/mol
* Diagnosis of T2D for at least 12 months
* General Practitioner responsible for diabetes treatment
* Residence in Hjørring, Morsø, Jammerbugt, or Rebild municipality
* Ability and willingness to use a smartphone/tablet along with the other devices to be used in the trial
* Signed informed consent
* Ability to understand and read Danish

Exclusion Criteria:

* Pregnancy or breastfeeding
* Insulin treatment
* Prednisolone treatment
* Severe diabetes complications such as severe neuropathy or nephropathy (dialysis treatment)
* Participation in diabetes rehabilitation courses
* Participation in other intervention trials
* Terms that, in the opinion of the sub-investigator or investigator, render the participant unfit to conduct the trial, including lack of understanding of the trial or lack of physical or cognitive ability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Experiences with and acceptability of intervention design(s) | 3 months
  Qualitative interviews will be conducted with selected participants and HCPs to gain deeper insight into the participants and HCPs' experiences and acceptability with the two different telemonitoring intervention designs and the trial procedures.

SECONDARY OUTCOMES:
Feasibility of the recruitment assessment 1 | 1 month
  Number (whole) of people agreeing to receive participant information letter about the study.
Feasibility of the recruitment assessment 2 | 1 month
  Proportion (percentage) of people agreeing to receive participant information letter about the study.
Feasibility of the recruitment assessment 3 | 1 month
  Number (whole) of eligible participants who agree to participate.
Feasibility of the recruitment assessment 4 | 1 month
  Proportion (percentage) of eligible participants who agree to participate.
Feasibility of the recruitment assessment 5 | 1 month
  Potential inequalities regarding recruitment feasibility assessed by comparing those who accepted participation to those who declined with respect to demographic data on age (years), sex (m/f/other), ethnicity (danish/other western/not western), municipality, setting (health care center versus home health care setting), and HbA1c levels (mmol/L).
Retention assessment 1 | 3 months
  Number (whole) of participants withdrawing from the trial.
Retention assessment 2 | 3 months
  Proportion (percentage) of participants withdrawing from the trial.
Retention assessment 3 | 3 months
  Timepoint(s) for withdrawal.
Retention assessment 4 | 3 months
  Reasons of discontinuation of the trial.
Retention assessment 5 | 3 months
  Potential inequalities regarding retention feasibility assessed by comparing those who retented participation to those who withdrawal with respect to demographic data on age (years), sex (m/f/other), ethnicity (danish/other western/not western), municipality, setting (health care center versus home health care setting), and HbA1c levels (mmol/L).
Adherence to answering the questionnaire: Diabetes-related quality of life: The Problem Areas in Diabetes Questionnaire (PAID-5) | At baseline (T0) and 3 months (T1)
  The respons rate for PAID-5 at baseline and at 3 months, respectively.
Adherence to answering the questionnaire: Quality of Life: The Short Form 12 Questionnaire (SF-12v2) | At baseline (T0) and 3 months (T1)
  The respons rate for SF-12v2 at baseline and at 3 months, respectively.
Adherence to answering the questionnaire: Well-being: The World Health Organization Five Well-being Index (WHO-5) | At baseline (T0) and 3 months (T1)
  The respons rate for WHO-5 at baseline and at 3 months, respectively.
Adherence to answering the questionnaire: The Patient Activation Measure questionnaire (PAM) | At baseline (T0) and 3 months (T1)
  The respons rate for PAM at baseline and at 3 months, respectively.
Challenges in the blood sampling schedule | At baseline (T0), 3 months (T1), 6 months (T2) and 12 months (T3)
  Explore through qualitative interviews whether there are any analysis challenges or uncertainties in the clinical workflow with regard to the blood sampling schedule.
Adherence to the blood sampling schedule | At baseline (T0), 3 months (T1), 6 months (T2) and 12 months (T3)
  Number and proportion of the participants who completes the blood sampling at baseline, 3 months, 6 months, and 12 months, respectively.
Costs | 12 months
  Differences in direct intervention costs between the two alternatives. Resource categories are comprised of equipment and time spent on monitoring, time spent training patients in using the equipment, and potential additional training for community nurses. Resources will be evaluated as prices paid and hourly wages and represented as equivalent annual costs in 2023 prices.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vestergaard, PhD (and MD), Principal Investigator — Aalborg University Hospital and Steno Diabetes Center North Denmark; Sisse H Laursen, PhD, Study Chair — Aalborg University and Aalborg University Hospital; Stine Hangaard, PhD, Study Chair — Aalborg University and Steno Diabetes Center North Denmark
Locations (1):
- Steno Diabetes Center North Denmark, Aalborg, Denmark

REFERENCES:
- [Derived] Laursen SH, Giese IE, Udsen FW, Hejlesen OK, Barington PF, Ohrt M, Vestergaard P, Hangaard S. A telemonitoring intervention design for patients with poorly controlled type 2 diabetes: protocol for a feasibility study. Pilot Feasibility Stud. 2024 May 22;10(1):83. doi: 10.1186/s40814-024-01509-0. PMID 38778345